CLINICAL TRIAL: NCT03028181
Title: The Evaluation of Pro/Antioxidative Profile and Diagnostic Parameters in the Patients With Acute Pancreatitis
Brief Title: The Evaluation of Pro/Antioxidative Profile and Diagnostic Parameters in the Patients With Pancreatic Disease
Status: Completed | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Milena Ściskalska, Principal Investigator, Wroclaw Medical University
Other Study IDs: 896-000-57-79
Record Dates: First submitted 2017-01-13; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Acute Pancreatitis
Keywords: smoke; acute pancreatitis; pro/antioxidant status; pro-inflammatory factors; lipid profile; exocrine functions of pancreas
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The blood samples taking into tubes containing heparin, EDTA and serum clotting activator to obtain plasma, erythrocyte lysate and serum.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Control group non-exposed to tobacco smoking
- 2: Control group exposed to tobacco smoking
- 3: Patients with acute pancreatitis non-exposed to tobacco smoking
- 4: Patients with acute pancreatitis exposed to tobacco smoking

SUMMARY:
The study aims to assess and analyze some selected antioxidants and laboratory parameters during hospitalization of the patients with acute pancreatitis. It will allow to better understanding of the mechanisms of disease and the development of better diagnostic, treatment and monitoring.

It is an observational diagnostic study and does not involve any additional administration of medicinal substances, modification of treatment or dropping the use of routine methods of treatment of a disease. The study procedure includes detailed personal medical history as separate document like as a routine medical interview, and three times taking a small amount of venous blood (together about 15 ml), in the first, third, and seventh day of hospitalization (in the case of longer hospital treatment).

ELIGIBILITY:
Inclusion Criteria:

* The patients were classified into the group of patients with acute pancreatitis (AP) due to clinical symptoms (acute onset of a persistent, severe, epigastric pain with tenderness on palpation on physical examination), personal interview and clinical method used in the diagnosis of pancreatitis - laboratory tests (elevation in serum lipase or amylase to three times or greater than the upper limit of normal) and characteristic findings of acute pancreatitis on imaging (contrast-enhanced computed tomography (CT), magnetic resonance imaging (MRI) or transabdominal ultrasonography). In patients with characteristic abdominal pain and elevation in serum lipase or amylase to three times or greater than the upper limit of normal, no imaging was required to establish the diagnosis of acute pancreatitis. In patients with abdominal pain that was not characteristic for acute pancreatitis or serum amylase or lipase levels that were less than three times the upper limit of normal, or in whom the diagnosis was uncertain, the investigators performed abdominal imaging with a contrast-enhanced abdominal CT scan to establish the diagnosis of acute pancreatitis and to exclude other causes of acute abdominal pain. In patients with severe contrast allergy or renal failure, the investigators performed an abdominal MRI without gadolinium.
* The volunteers classified as healthy based on the research conducted by clinicians of primary medical care (control group)

Exclusion Criteria:

* other accompanied diseases than acute pancreatitis (the patients groups)
* Individuals of the control group with diagnosed disease as well as alcohol and drugs abusers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. The healthy volunteers classified as a control group based on the research conducted by clinicians of primary medical care, divided on smokers and non-smokers.
  2. The patients classified into the group of patients with acute pancreatitis, divided on smokers and non-smokers.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pro-inflammatory effect of tobacco smoke exposure measured by hsCRP concentration in the blood of patients with acute pancreatitis | 3 weeks
Pro-inflammatory effect of tobacco smoke exposure measured by Interleukin-6 concentration in the blood of patients with acute pancreatitis | 2 weeks

SECONDARY OUTCOMES:
The estimation of antioxidant status measured by the activities of antioxidant enzymes in the blood | 12 months
The estimation of antioxidant status measured by small molecular antioxidants concentration in the blood | 3 months
The estimation of prooxidant status measured by the concentration of lipids peroxidation products in the blood | 2 months
The estimation of prooxidant status measured by the concentration of advanced oxidation protein products in the blood | 1 months

OTHER OUTCOMES:
The estimation of the concentration of vascular endothelium damage marker (endothelin) in the blood | 3 months
The estimation of the concentration of total cholesterol in the blood | 3 weeks
The estimation of the concentration of triglycerides in the blood | 3 weeks
The estimation of the concentration of low-density lipoprotein (LDL) in the blood | 3 months
The estimation of the concentration of high-density lipoprotein (HDL) in the blood | 3 weeks
The estimation of endocrine functions of pancreas measured by the concentration of insulin in the blood | 2 months
The estimation of endocrine functions of pancreas measured by the concentration of glucagon in the blood | 1 month
The estimation of endocrine functions of pancreas measured by the concentration of pancreatic polypeptide in the blood | 1 month
The estimation of endocrine functions of pancreas measured by the concentration of somatostatin in the blood | 1 month
The estimation of endocrine functions of pancreas measured by the concentration of ghrelin in the blood | 2 weeks
The estimation of exocrine functions of pancreas measured by the activity of amylase and lipase in the blood | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Halina Milnerowicz, Prof., Study Chair — Wroclaw Medical University, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No